CLINICAL TRIAL: NCT03896126
Title: Instantaneous Measures of Autonomic Nervous System Responses to Gastrointestinal Challenges
Brief Title: GI-Challenge Study for Gastroparesis Patients and Healthy Controls
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to technical issues with the ANSAR equipment, lack of research personnel caused by COVID-19 restrictions imposed at our site, and recent departure of the PI and study chair from our research institute.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Linda Nguyen, Clinical Professor - Medicine/Gastroenterology and Hepatology, Stanford University
Other Study IDs: 44258
Record Dates: First submitted 2019-03-15; First posted 2019-03-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Gastroparesis
Keywords: Healthy Control; Diabetic Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Gastroparesis Patients: 20 gastroparesis patient ages 20-49
  Interventions: Other: Observational
- Healthy Controls: 40 healthy controls ages 20-49
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — There is no intervention. This is an observational study attempting to establish parameters of normal and abnormal vagal tone in healthy control and gastroparesis patients, as there is currently no metric to determine what dose of vagal stimulation is required to treat gastroparesis.

SUMMARY:
Gastroparesis Patients and Healthy Controls ages 20-49 will be asked to participate in an observational study measuring vagal activity following food ingestion in order to establish parameters of autonomic nerve/vagal function in healthy human subjects compared to those with gastroparesis. Information generated from this study may be used in the future to establish what is normal and abnormal enteric vagal tone and how much vagal nerve stimulation treatment may be required to help patients with gastroparesis.

DETAILED DESCRIPTION:
Impaired function of the vagus nerve has been documented in many chronic diseases such as diabetes, heart disease, and chronic pain, as well as gastrointestinal diseases such as irritable bowel syndrome, inflammatory bowel disease, and delayed stomach emptying (gastroparesis).

Current technology only allows for measurement of vagal nerve activity that regulates the heart and diagnostic tests focus specifically on cardiac vagal activity. Measuring vagal nerve activity as it pertains to the gastrointestinal system is an unmet medical need. Its importance will continue to grow since vagal nerve stimulation is being used increasingly in a myriad of different diseases, and currently there is no way of knowing if patients are getting too little or too much stimulation.

In this study, the gastrointestinal vagus nerve will be activated using normal stimulants like food ingestion and vagal activity will be measured using current non-invasive technology. Patients with gastroparesis and healthy controls will be asked to come in fasting, fill out surveys, and complete eating challenges while being connected to an autonomic function testing machine. Exploratory outcomes will also be measured - Participants will be connected to a Peripheral Intravenous Line in order to collect four vials of blood throughout the two hour clinic visit so that hormonal changes can be studied. Also, exploratory non-invasive electrogastrograms will be recorded remotely both during the autonomic function test and for three consecutive days as participants go about their daily lives.

The investigators' goal is to establish a protocol for measuring gastrointestinal evoked vagal activity and correlating activity with digestive function in both healthy people and gastroparesis patients.

ELIGIBILITY:
Inclusion Criteria

1. Male or female.
2. Age 20-49 years old.
3. Healthy volunteer or established diagnosis of idiopathic gastroparesis as per AGA (American Gastroenterology Association) guidelines.
4. Participant is capable of giving informed consent.
5. Gastroparesis patients must be on stable doses of medications for gastroparesis for preceding 4 weeks prior to enrollment (including cholinergics, anti-cholinergics, dopamine and serotonin receptor agonists/antagonists, motility agents, neuromodulators, herbals).

Exclusion criteria.

1. Diagnosis of systemic autonomic nerve dysfunction (i.e. POTS, CAN).
2. Surgical-related gastroparesis
3. Extrinsic myopathy or neuropathy causing gastroparesis.
4. Use of narcotic pain medications in the preceding 2 weeks of study enrollment.
5. Patients with enteric feeding tubes or requiring parenteral nutrition.
6. Patients with severe disease flare requiring hospitalization or frequent emergency room visits (last within 3 months or less of enrollment).
7. Untreated significant depression or suicidal thoughts.
8. Pregnant or breast-feeding women.
9. History of gastric pacemaker implantation.
10. Patients with prior gastric surgery, including fundoplication, partial/total gastrectomy, pyloroplasty, or gastric bypass.
11. Patients with implantable electronic devices.
12. Dairy, wheat, or egg allergy/intolerance.
13. Allergy to commercial clinical adhesive for EKG stickers.
14. Non-English speaker and/or hearing impaired (as participants need to follow English verbal commands and cues for the experiment).

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 Patients (20 Gastroparesis and 40 Controls) between the ages of 20-49.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Determination of sympathovagal score, a measure of cardiac autonomic activity, following digestive challenges in healthy volunteers using the FDA-approved ANSAR ANX 3.0 Autonomic Nervous System (ANS) Monitoring System. | Single two hour visit
  The ANSAR computes sympathovagal score by collecting sympathetic low frequency area (LFa) and parasympathetic respiratory frequency area (RFa) data (both measured as beats per minute squared, or BPM2) and calculating the ratio of these two complementary measures of the autonomic nervous system (LFa/RFa) to arrive at one aggregated score.
Determination of sympathovagal score following digestive challenges in gastroparesis patients using the ANSAR ANX 3.0 ANS Monitoring System and comparison to healthy volunteers. | Single two hour visit
  The ANSAR computes sympathovagal score by collecting sympathetic low frequency area (LFa) and parasympathetic respiratory frequency area (RFa) data (both measured as beats per minute squared, or BPM2) and calculating the ratio of these two complementary measures of the autonomic nervous system (LFa/RFa) to arrive at one aggregated score.
Correlation of sympathovagal score, a measure of cardiac autonomic activity, with gastroparesis disease severity. | Single two hour visit
  To determine if sympathovagal scores correlate with gastroparesis clinical disease severity using standardized GI symptom scoring - the Gastroparesis Cardinal Symptom Index consists of 10 questions that rate gastroparesis symptoms on a scale of 1 - 6 from "none" to "very severe".

CONTACTS AND LOCATIONS:
Overall Officials: Andres C Gottfried Blackmore, MD, PhD, Principal Investigator — Stanford University; Linda Nguyen, MD, Study Chair — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No